CLINICAL TRIAL: NCT05363046
Title: A Multi-center, Noninterventional Study Evaluating Variability, Reliability, and Compliance for the Parkinson's Disease Diary
Brief Title: Noninterventional Study Evaluating Parkinson's Disease Diary Use
Status: Active, not recruiting | Type: Observational
Sponsor: BlueRock Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: BRT-DA01-NIS-001
Record Dates: First submitted 2022-05-03; First posted 2022-05-05 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Participants will complete the PD diary on 3 consecutive days in 1 week.
- Group B: Participants will complete the PD diary on 2 consecutive days in each of 2 consecutive weeks.

SUMMARY:
This study aims to evaluate the impact of the frequency of assessments on the variability over time, reliability, and compliance for the Parkinson's disease (PD) diary in patients with PD in whom medications do not provide adequate control of symptoms.

DETAILED DESCRIPTION:
This is a global, multi-center, noninterventional study of patients with PD aged ≥39 to ≤70 years under standard-of-care treatment that will enroll a minimum of approximately 150 participants and up to 400 participants. Participants will be assigned (1:1) to complete the PD diary either on 3 consecutive days in 1 week (Group A) or 2 consecutive days in each of 2 consecutive weeks (Group B) for a given study visit. During the study, data are collected on motor function, quality of life, and use of PD medications at Baseline and at 3, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria

* ≥39 to ≤70 years of age at signing of informed consent
* Diagnosis of clinically established PD as defined by the Movement Disorder Society (MDS) Clinical Diagnostic Criteria for PD
* Marked levodopa responsiveness at screening per investigator's judgment (eg, an estimated ≥30% improvement of MDS-UPDRS Part III score in the off-medication versus on-medication state)
* A minimum of 3 years and a maximum of 10 years from time of PD diagnosis to the date of screening
* Receiving optimized and stable PD medical therapy for ≥1 month prior to screening or demonstrated intolerance to PD medications per investigator's judgment in agreement with the medical monitor
* ≥2 hours of average daily OFF-time assessed within 3 months of screening by PD diary or per investigator's judgment
* Hoehn and Yahr Stage of 1 to 3 while on PD medication assessed within 3 months of screening or at screening
* Normal cognition as determined by the investigator after review of relevant testing (eg, Montreal Cognitive Assessment score of ≥26, or ≥22 if no significant cognitive impairment as determined by neuropsychological testing)

Exclusion Criteria:

* PD with risk of recurrent falls or only tremor-based symptoms
* Diagnosis of primary mitochondrial disorder, epilepsy, stroke, multiple sclerosis, or clinical features suggestive of a neurodegenerative disease other than PD such as Alzheimer's disease
* Any available evidence inconsistent with dopamine deficiency (eg, 18F-DOPA positron emission tomography [PET] or dopamine transporter single-photon emission computed tomography [DAT-SPECT] imaging if performed)
* Moderately severe dyskinesia per investigator's judgment
* Receiving dopamine receptor-blocking agents, including typical neuroleptics, prochlorperazine, and metoclopramide at the time of screening or within 3 months prior to screening
* Treatment with intrajejunal or subcutaneous infusion therapies for PD within 2 months of screening
* History of gene therapy or cell therapy
* Prior surgical or radiation therapy to the brain, including deep brain stimulation and lesion therapy, or prior history of intradural spinal cord surgery
* Receipt of another investigational therapy or device within 2 years of screening unless approved by the medical monitor

Ages: 39 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients whose medications do not provide adequate control of their symptoms.
Sampling Method: Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Good ON-time as measured by the PD Diary. | Baseline, 3, 6, 12, 18 and 24 months.
  Standard deviation of change in ON-time without troublesome dyskinesia (Good ON-time) as measured by the PD diary.
Individual participant variability for ON-time without troublesome dyskinesia (Good ON-time) as measured by the PD diary. | Baseline, 3, 6, 12, 18 and 24 months.
  Within-subject coefficient of variation for ON-time without troublesome dyskinesia (Good ON-time) as measured by the PD diary.
Proportion of valid PD Diaries. | Baseline, 3, 6, 12, 18 and 24 months.
  Proportion of valid PD Diaries.

CONTACTS AND LOCATIONS:
Locations (34):
- United States (16):
  - Mayo Clinic Neurology, Scottsdale, Arizona
  - David Geffen School of Medicine University of California Los Angeles, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of Colorado, Aurora, Colorado
  - Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Miami Health System, Miami, Florida
  - Parkinson's Disease and Movement Disorders Center at Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Mount Sinai West, New York, New York
  - Weill Cornell Medicine - New York Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Evergreen Health Medical Center, Kirkland, Washington
- Toronto Western Hospital, Toronto, Ontario, Canada
- Germany (8):
  - Dkd Wiesbaden, Wolfach, Baden-Wurttemberg
  - Klinikum der Universität München - Campus Grosshadern, Munich, Bavaria
  - Technischen Universitaet Muenchen (TUM), Munich, Bavaria
  - Universitätsklinikum Würzburg - Medizinische Klinik, Würzburg, Bavaria
  - Klinik und Poliklinik für Neurologie am Standort Marburg, Marburg, Hesse
  - Universitaetsklinikum Duesseldorf AöR, Düsseldorf
  - Universitätsmedizin Rostock, Rostock
  - University Hospital Tuebingen, Tübingen
- Italy (4):
  - AOU Ospedali Riuniti Umberto I - G.M. Lancisi - G. Salesi, Ancona
  - Azienda Ospedale Università Padova, Padua
  - IRCCS San Raffaele Pisana, Rome
  - AOU OO.RR. San Giovanni di Dio Ruggi d'Aragona, Salerno
- Spain (5):
  - Hospital San Juan de Dios, Santurtzi, Bilbao
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Complexo Hospitalario de Pontevedra (CHOP), Pontevedra
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No